CLINICAL TRIAL: NCT01002131
Title: Exact Three-dimensional Localisation of Impacted and Supernumerary Teeth by Cone Beam Computer Tomography
Brief Title: Exact Localisation of Impacted and Supernumerary Teeth by Cone Beam Computer Tomography
Status: Completed | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 19236
Record Dates: First submitted 2009-10-26; First posted 2009-10-27 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Impacted Teeth
Keywords: Digital Volume Tomography; Cone Beam CT; impacted and supernumerary teeth; dental and maxillofacial radiology
MeSH Terms: conditions — Tooth, Impacted; Tooth, Supernumerary

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Digital Volume tomography: three-dimensional digital imaging using cone beam tomography (CBCT)
  Interventions: Device: CBCT

INTERVENTIONS:
Device: CBCT — Cone Beam Computer Tomography. 3D-imaging Digital Volume Tomography, compared with gold standard intraoperative findings.
  Other Names: Cone Beam Tomography; i-Cat device; digital volume tomography (DVT)

SUMMARY:
The purpose of this investigation is an exact preoperative 3D-localisation of impacted and supernumerary teeth in the maxilla using Cone Beam Computer Tomography

DETAILED DESCRIPTION:
An exact localisation of impacted teeth is often difficult to assume by using conventional radiological techniques like OPT or dental films. In contrast to these two-dimensional imaging methods the Cone Beam Computer Tomography (CBCT) respectively the Digital Volume Tomography (DVT) offers a three-dimensional imaging of the maxillofacial region, providing the opportunity to study objectives in all standard plans with 3D-reconstruction in multisection views.

A preoperative radiological investigation using CBCT on patients who are supposed to undergo surgery for impacted and supernumerary teeth in the frontal maxilla shall clarify the certainty and safeness of this 3D-imaging method. Therefore a comparison between the findings on the CBCT, on eventually former conventional x-rays and the intraoperative finding as gold standard is done.

ELIGIBILITY:
Inclusion Criteria:

* supernumerary and impacted teeth in the maxilla (wisdom teeth excluded)
* need for surgical removement
* uncertain clinical and conventional radiological finding

Exclusion Criteria:

* refused approval
* CBCT not practicable

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients at the St.Olavs University Hospital with impacted and supernummerary teeth in the maxilla who are scheduled to have surgery
Sampling Method: Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2007-05 (Actual); Primary Completion 2009-04 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
exact localisation of impacted teeth | preoperative and under surgery
  Cone Beam Computer Tomography, vs gold standard intraoperative finding

CONTACTS AND LOCATIONS:
Overall Officials: Christoph M Ziegler, Professor, Study Director — NTNU / St.Olavs Hospital; Thomas R Klimowicz, PhD, Principal Investigator — St. Olavs Hospital
Locations (1):
- St Olavs Hospital, Trondheim, Norway

REFERENCES:
- [Result] Ziegler CM, Klimowicz TR. A comparison between various radiological techniques in the localization and analysis of impacted and supernumerary teeth. Indian J Dent Res. 2013 May-Jun;24(3):336-41. doi: 10.4103/0970-9290.117998. PMID 24025881